CLINICAL TRIAL: NCT02590679
Title: Multi-center Trial of Percutaneous Pulmonary Valve Implantation Using Venus-P Valve for Patients With Severe Pulmonary Regurgitation and Native Right Ventricular Outflow Tract After Previous Surgical Repair
Brief Title: Multi-center Trial of Percutaneous Pulmonary Valve Implantation With Venus-p
Acronym: Venus-P
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other); Huaxi Hospital (Other); Shanghai Chest Hospital (Other); Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPVI-2013
Record Dates: First submitted 2015-10-15; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Pulmonary Regurgitation; Tetralogy of Fallot
MeSH Terms: conditions — Pulmonary Valve Insufficiency; Tetralogy of Fallot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRAS (Experimental): pulmonary regurgitation after surgical repair of congenital right ventricular outflow tract
  Interventions: Device: Venues-P Valve

INTERVENTIONS:
Device: Venues-P Valve — a Novel Self-Expanding Percutaneous Stent-Valve in the Native Right Ventricular Outflow Tract

SUMMARY:
Venus-P Valve (Venus Medtech, Shanghai, China) is the first self-expandable interventional Pulmonary Valve, which is composed of a Nitinol multilevel support frame with a tri-leaflet porcine pericardial tissue valve, and a 14-22 Fr delivery catheter. The purpose of the multi-center trial is to evaluate the safety and efficacy of the Venus-P Valve for percutaneous pulmonary valve implantation (PPVI) in patients pulmonary regurgitation and native right ventricular outflow tract (RVOT) after surgical repair of RVOT.

DETAILED DESCRIPTION:
Clinical experience to date with transcatheter pulmonary valve replacement has been limited to two balloon expandable systems, namely the Melody Valve (Medtronic Inc, Minneapolis, MN) and the Sapien valve (Edwards Lifesciences, Irvine, CA). Both valves have undergone clinical trials with good medium-term valve durability. Although both the Melody and the Sapien valves have been used in native outflow tracts with good success , limitations to the extended application of these valves have generally centered on the maximum diameter of the RVOT. Indeed in the majority of patients requiring pulmonary valve replacement (PVR), these balloon expandable systems are not large enough to maintain stable valve position within the dilated native RVOT.Therefore more recent efforts have concentrated on a self-expanding system to provide valve competence despite significant dilation of the native RVOT.

Venus-P Valve (Venus Medtech, Shanghai, China) is the first self-expandable interventional Pulmonary Valve, which is composed of a Nitinol multilevel support frame with a tri-leaflet porcine pericardial tissue valve, and a 14-22 Fr delivery catheter. The purpose of the trial is to evaluate the safety and efficacy of the Venus-P Valve for PPVI in patients pulmonary regurgitation and native RVOT after surgical repair of RVOT.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe pulmonary regurgitation after surgical repair of congenital right ventricular outflow tract obstruction with trans-annulus or RVOT patch;
2. right ventricular diastolic volume index: 130-160 mL/m2 measured by isotopic examination or cardiac MRI measurements;
3. Age: ≥10 years and ≤60 years;
4. Weight ≥18 Kg;
5. Pulmonary annulus : 14- 31 mm;
6. RVOT length ≥20mm ;
7. Signing the informed consent;
8. Any of the following conditions: ① symptomatic, ②progressive RV systolic dysfunction, ③ progressive tricuspid regurgitation (at least moderate), ④ RVOT obstruction with RV systolic pressure ≥80 mmHg, ⑤ Sustained atrial/ventricular arrhythmias.

Exclusion Criteria:

1. Pre-existing pulmonary artery stenosis or artificial pulmonary valve at any position;
2. Severe chest wall deformity (funnel chest, etc.);
3. Acute uncompensated heart failure;
4. Active infection or endocarditis requiring antibiotic therapy;
5. Leukopenia (white blood cell <3000 mm3);
6. Acute or chronic anemia (hemoglobin <9 g/L);
7. Platelet counts <10000 /mm3;
8. Impossibly of delivering Venus-P to RVOT as judged by researcher s before procedure;
9. Known allergy to aspirin or heparin;
10. Positive urine or serum pregnancy test in female subjects.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-07 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
right ventricular end diastolic volume index | 6 months

SECONDARY OUTCOMES:
Incidence of adverse cardiovascular events | 48 hours
  death, severe arrhythmia, pericardial tamponade, emergency surgery, RVOT rupture, pulmonary artery perforation, cardiac shock, endocarditis, bleeding , and other complications caused by procedure
Incidence of deaths or strokes | 12 months
  All cause deaths (cardiac death, and non cardiac death) or strokes
pulmonary pressure gradient | 1,3,6,12 months
  Max pressure gradient (PG)
grade of pulmonary regurgitation | 1,3,6,12 months
New York Heart Association (NYHA) class | 1,3,6,12 months
6 minutes walk distance | 1,3,6,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, M.D., Study Chair — Fudan University
Locations (3):
- China (3):
  - Zhongshan Hopital of Fudan University, Shanghai, Shanghai Municipality
  - Beijing Fuwai Hospital, Beijing
  - Shanghai Chest Hospital, Shanghai

REFERENCES:
- [Result] Cao QL, Kenny D, Zhou D, Pan W, Guan L, Ge J, Hijazi ZM. Early clinical experience with a novel self-expanding percutaneous stent-valve in the native right ventricular outflow tract. Catheter Cardiovasc Interv. 2014 Dec 1;84(7):1131-7. doi: 10.1002/ccd.25544. Epub 2014 May 28. PMID 24824357